CLINICAL TRIAL: NCT04023006
Title: An Observational Clinical Case Series Study to Assess Fit and Quality of Full Dentures
Brief Title: An Observational Clinical Case Series Study to Assess Fit and Quality of Full Dentures Fabricated by AM
Status: Terminated | Type: Observational
Why Stopped: No usable data were obtained. Therefore, the study was terminated.
Sponsor: Dentsply International (Industry)
Responsible Party: Sponsor
Organization: Dentsply Sirona Inc. (Industry)
Other Study IDs: PRPA 22901 / CR 02
Record Dates: First submitted 2019-07-12; First posted 2019-07-17 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Mouth, Edentulous
Keywords: Denture
MeSH Terms: conditions — Mouth, Edentulous

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Edentulous Patients: The investigational device is part of a treatment concept for edentulous patients of all ages, gender and races. The incidence for tooth loss has not declined over years, and the prevalence for edentulism is significantly higher for adults 50 years and older. For this descriptive two-part survey, no minimum number of patients is defined, but to achieve a reasonable subject number, a minimum of five (5) patients will be enrolled, i.e. 10 dentures will be fabricated within this study.
  Interventions: Device: Removable prostheses

INTERVENTIONS:
Device: Removable prostheses — Full dentures created by Additive manufacturing (Carbon Printers)
  Other Names: Lucitone 3D print resin dentures

SUMMARY:
This observational clinical case series investigation will be conducted on approximately five (5) enrolled subjects at one (1) site in the US. Treatment of subjects encompasses all steps to fabricate new dentures for maxilla and/or mandible. The subjects will be followed 7-10 days after final delivery of the denture

DETAILED DESCRIPTION:
This investigation is undertaken to evaluate the workflow and concomitant products to create full dentures by using additive manufacturing (AM) technology, i.e. Digital Light Processing™ Technology (Carbon 3D) to restore fully edentulous jaws. The assessment includes quality of materials provided by Dentsply Sirona Lab by using printers for AM (M series, Carbon 3D 1089 Mills Way, Redwood City, CA 94063). This assessment will be done by clinical review of the AM dentures on fit and quality. In addition, the evaluation includes a patient survey to assess current dentures and the new AM dentures with a subjective comparison of both.

The target subjects are male or female, 18 years and older with the need of a full denture in one or both jaws, being completely edentulous. The newly fabricated denture is to replace an existing full denture. For this descriptive study, no minimum number of patients is defined, but to achieve a reasonable subject number, a minimum of five (5) and a maximum of ten (10) patients will be enrolled, i.e. ten to twenty (10-20) denture arches will be fabricated within this study.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years or older.
* Subject has given written consent to participate in the trial.
* Subject is in good general health.
* Subject requires a new removable full denture for both jaws.
* Subject is completely edentulous in the maxilla and mandible.
* Subject is already wearing a full denture in the maxilla and mandible.
* Subject is willing to undergo dental treatment to receive a new full denture for both jaws.
* Subject confirms availability for treatment and all indicated follow-up visits.

Exclusion Criteria:

* Subject is younger than 18 years.
* Subject is pregnant.
* Subject has disabilities that do not allow a regular dental treatment.
* Subject with some systemic medical complications that cause difficulty in impression taking or judging occlusion of device.
* Subject is currently participating in another study.
* Subject has an allergic history regarding materials used in this trial.
* Subject with xerostomia/ dry-mouth syndrome.
* Lack of compliance is expected.
* Those subjects who cannot provide informed consent for any reason
* Acute stomatitis.
* Status after tumor treatment in head-neck region (removal, radiotherapy).
* Acute cancer.
* Incomplete hard and/or soft tissue in the oral cavity.
* Muscle and/or nerve damage in the head-neck region.
* Insufficient vertical height and/or insufficient mouth opening.
* Resilient hyperplastic mucosa ("flappy ridges").
* Bruxism.
* Insufficient oral hygiene. The existing dentures should have no visible calculus.
* Previously enrolled in the present investigation.
* Involvement in the planning and conduct of the clinical investigation. (applies to all Dentsply Sirona & Carbon 3D staff, investigational site staff staff and third party vendor).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigational device is part of a treatment concept for edentulous patients of all ages, gender and races. The incidence for tooth loss has not declined over years, and the prevalence for edentulism is significantly higher for adults 50 years and older. For this descriptive two-part survey, no minimum number of patients is defined, but to achieve a reasonable subject number, a minimum of five (5) patients will be enrolled, i.e. 10 dentures will be fabricated within this study.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Assessment of the fit of the denture | At Final Placement of Denture, through study completion, an average of one month
  A questionnaire of assessment of fit by ranking, in comparison to the previous denture, using a Likert Scale from a minimum of 5 to a maximum of 1.
  Much worse (5) Worse (4) Same (3) Better (2) Much better (1)

SECONDARY OUTCOMES:
Aesthetics of dentures | At Final Placement of Denture,through study completion, an average of one month
  A questionnaire of assessment of aesthetics by ranking, in comparison to the previous denture, using a Likert Scale from a minimum of 5 to a maximum of 1.
  Much worse (5) Worse (4) Same (3) Better (2) Much better (1)
Function of dentures | At Final Placement of Denture,through study completion, an average of 1 month
  A questionnaire of assessment of function by ranking, in comparison to the previous denture, using a Likert Scale from a minimum of 5 to a maximum of 1.
  Much worse (5) Worse (4) Same (3) Better (2) Much better (1)
Dentist's satisfaction with treatment: questionnaire | At Final Placement of Denture, through study completion, an average of 1 month
  A questionnaire of assessment of satisfactions of treatment by ranking, in comparison to the previous placed denture, using a Likert Scale from a minimum of 5 to a maximum of 1.
  Much worse (5) Worse (4) Same (3) Better (2) Much better (1)

CONTACTS AND LOCATIONS:
Locations (1):
- Boston University Goldman School of Dental MEdicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Celebic A, Knezovic-Zlataric D, Papic M, Carek V, Baucic I, Stipetic J. Factors related to patient satisfaction with complete denture therapy. J Gerontol A Biol Sci Med Sci. 2003 Oct;58(10):M948-53. doi: 10.1093/gerona/58.10.m948. PMID 14570864
- [Background] Schwindling FS, Bomicke W, Hassel AJ, Rammelsberg P, Stober T. Randomized clinical evaluation of a light-cured base material for complete dentures. Clin Oral Investig. 2014;18(5):1457-65. doi: 10.1007/s00784-013-1110-4. Epub 2013 Sep 21. PMID 24057919